CLINICAL TRIAL: NCT06507566
Title: Phase 1 Study Evaluating Technologies for Point-of-Care Blood Collections in Support of Decentralized Outpatient Assessments in Pandemic and Clinical Trial Settings
Brief Title: Evaluating Technologies for Point-of-Care Blood Collections by Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Collaborators: ICON Government and Public Health Solutions, Inc (Unknown); Joint Program Executive Office Chemical, Biological, Radiological, and Nuclear Defense Enabling Biotechnologies (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 5309/0024
Record Dates: First submitted 2024-06-24; First posted 2024-07-18 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Tasso, Tasso+

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cohort A (Active Comparator): Samples centrifuged/aliquoted after arrival at central lab.
  Interventions: Device: Tasso+™
- Cohort B (Active Comparator): Samples centrifuged/aliquoted at collection Site before shipment to central lab.
  Interventions: Device: Tasso+™

INTERVENTIONS:
Device: Tasso+™ — The Tasso+™ blood collection kit is a collection device (called the Tasso+™) and a capillary collection tube that allows for the storage of the blood in a liquid format in different matrices.

SUMMARY:
A study evaluating technologies for point-of-care use in clinical trials.

DETAILED DESCRIPTION:
A study evaluating the Tasso+ blood collection device that enables the safe and convenient collection of blood by a lay person (eg, patient or study participant) under the supervision of an Health Care Provider.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults (18 years of age or older, inclusive), at the time of informed consent. Participants who are deemed pregnant by urine pregnancy test at Screening remain eligible.
* Able to understand and willing to provide informed consent and able to comply with the study procedures and restrictions.
* Participant considered healthy or in well-compensated health according to medical history, concomitant medications, and physical examination (including vital signs).

Exclusion Criteria:

* Medical history, or physical examination (including vital signs) findings, that suggest to the Investigator that the participant has undiagnosed or untreated medical condition(s) that could confound the AE evaluation and thereby undermine the study objectives.
* Any known medical history of infection with HIV (CD4<200 and/or detectable viral load within the prior 3 months), hepatitis B (positive HBsAg), or hepatitis C (positive hepatitis C virus antibody).
* Chronic illness for which a participant's immune system is suspected by the Investigator to be impaired or altered, such as cancer, autoimmune conditions, and diabetes.
* Participation in another investigational study within 30 days of time of consent or plans to do so during the course of this study.
* Large tattoos or skin eruptions overlying either of the deltoid muscles that could confound the monitoring for local reactogenicity following Tasso+™ administrations.
* Use of systemic immunomodulatory therapy, including oral corticosteroids, within the past 6 months; or planned use of medications or nutritional supplements known to or which potentially could affect organ function within 30 days prior to screening until end of study.
* Acute illness within 14 days prior to device use unless it is determined by the Investigator that the illness is mild in severity and unlikely to progress.
* Of limited legal capacity.
* Any condition (including suspected alcohol- or drug-related addiction) that precludes adequate understanding, cooperation, and/or compliance with study procedures or any condition that could pose a risk to the participant's safety per Investigator judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-10-29 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Victor Salib, Riverside, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 134 | 66
Completed | 120 | 57
Not Completed | 14 | 9
Not completed — Lost to Follow-up | 9 | 7
Not completed — Withdrawal by Subject | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 134 | 66 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (17.22) | 40.6 (15.79) | 41.8 (16.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 42 | 124
  Male | 52 | 24 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59 | 31 | 90
  Not Hispanic or Latino | 74 | 34 | 108
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 16 | 9 | 25
  White | 110 | 54 | 164
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Weight [Mean (Standard Deviation); unit: kg] | 85.67 (23.99) | 83.16 (19.83) | 84.84 (22.68)
Height [Mean (Standard Deviation); unit: m] | 1.69 (0.11) | 1.69 (0.1) | 1.69 (0.11)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.03 (7.7) | 29.15 (6.84) | 29.74 (7.42)

OUTCOME MEASURES:

1. Primary Outcome: Assess the Sample Integrity of Tasso+™
Description: Percentage of overall Tasso+™/serum separator tube (SST) samples collected that are with adequate volume and without moderate or gross hemolysis
Time Frame: Day 1
Population: Per the SAP, the full analysis set is defined as all participants who administered Tasso+™ either in a site-supervised, proctor supported, or unsupported setting (regardless of cohort). This analysis set will be the primary set used for analyses/summaries of the primary endpoint, as well as for secondary endpoints of seroconversion.
Measure: Number; unit: percentage of samples
Units Other Than Participants: Samples
Groups:
- Total: All subjects with samples centrifuged/aliquoted after arrival at central lab and samples centrifuged/aliquoted at collection site before shipment to central lab.
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 123 | 63 | 186
Number analyzed (Samples) | 123 | 63 | 186
percentage of samples | 23.1 | 75.8 | 40.5

2. Primary Outcome: Assess the Sample Integrity of Tasso+™
Description: as for outcome 1
Time Frame: Day 29
Population: Per the SAP, the full analysis set is defined as all participants who administered Tasso+™ either in a site-supervised, proctor supported, or unsupported setting (regardless of cohort). This analysis set will be the primary set used for analyses/summaries of the primary endpoint, as well as for secondary endpoints of seroconversion. The analysis population in the Day 29 endpoints includes all subjects regardless of cohort.
Measure: Number; unit: percentage of samples
Units Other Than Participants: samples
Arm/Group | Total
Number analyzed (Participants) | 163
Number analyzed (samples) | 163
percentage of samples | 29.5

3. Primary Outcome: Assess the Sample Integrity of Tasso+™
Description: as for outcome 1
Time Frame: Day 57
Population: Per the SAP, the full analysis set is defined as all participants who administered Tasso+™ either in a site-supervised, proctor supported, or unsupported setting (regardless of cohort). This analysis set will be the primary set used for analyses/summaries of the primary endpoint, as well as for secondary endpoints of seroconversion. The analysis population in the Day 57 endpoints includes all subjects regardless of cohort.
Measure: Number; unit: percentage of samples
Units Other Than Participants: samples
Arm/Group | Total
Number analyzed (Participants) | 140
Number analyzed (samples) | 140
percentage of samples | 28

4. Primary Outcome: Assess the Sample Integrity of Tasso+™
Description: Percentage of overall Tasso+™/ ethylenediaminetetraacetic acid (EDTA) samples collected that are with adequate volume, without moderate or gross hemolysis, and without clotting
Time Frame: Day 1
Population: as for outcome 1
Measure: Number; unit: percentage of samples
Units Other Than Participants: samples
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 124 | 65 | 189
Number analyzed (samples) | 124 | 65 | 189
percentage of samples | 2.2 | 43.9 | 16.0

5. Primary Outcome: Assess the Sample Integrity of Tasso+™
Description: as for outcome 4
Time Frame: Day 29
Population: as for outcome 2
Measure: Number; unit: percentage of samples
Units Other Than Participants: samples
Arm/Group | Total
Number analyzed (Participants) | 159
Number analyzed (samples) | 159
percentage of samples | 2.5

6. Primary Outcome: Assess the Sample Integrity of Tasso+™
Description: as for outcome 4
Time Frame: Day 57
Population: as for outcome 3
Measure: Number; unit: percentage of samples
Units Other Than Participants: samples
Arm/Group | Total
Number analyzed (Participants) | 141
Number analyzed (samples) | 141
percentage of samples | 2.5

7. Primary Outcome: Assess the Testing Accuracy of Tasso+™
Description: Correlation of SARS-CoV-2 (positive for IgG antibody) serology between venipuncture and Tasso+™/SST or Tasso+™/EDTA samples for Cohort A
Time Frame: Day 1
Population: as for outcome 1
Measure: Number; unit: percentage of samples
Units Other Than Participants: samples
Arm/Group | Cohort A
Number analyzed (Participants) | 134
Number analyzed (samples) | 134
percentage of samples
  Venipuncture/(SST or EDTA) | 41.04
  Tasso+™/(SST or EDTA) | 41.79
Statistical Analysis 1: Comparison: Cohort A; Test type: Other — Pearson's correlation coefficient were computed to quantify the strength of the direction of the linear relationship between the venipuncture collection and the Tasso+™ collection at Day 1 for each cohort for SARS-CoV-2 serology. Contingency correlation coefficient was computed to estimate the extent of the relationship between the venipuncture collection and the Tasso+™ collection at Day 1 for each cohort for SARS-CoV-2 serology; Correlation contingency coefficient = 0.70

8. Primary Outcome: Assess the Testing Accuracy of Tasso+™
Description: Correlation of SARS-CoV-2 (positive for IgG antibody) serology between venipuncture and Tasso+™/SST or Tasso+™/EDTA samples for Cohort B
Time Frame: Day 1
Population: as for outcome 1
Measure: Number; unit: percentage of samples
Units Other Than Participants: samples
Arm/Group | Cohort B
Number analyzed (Participants) | 66
Number analyzed (samples) | 66
percentage of samples
  Venipuncture/(SST or EDTA) | 53.03
  Tasso+™/(SST or EDTA) | 46.97
Statistical Analysis 1: Comparison: Cohort B; Test type: Other — [test comment as in outcome 7, analysis 1]; Correlation Contingency Coefficient = 0.68

9. Primary Outcome: Assess the Testing Accuracy of Tasso+™ as Compared to Samples Collected Via Venipuncture for Sodium
Description: Correlation of sodium between venipuncture and Tasso+™/SST samples for each cohort
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Units Other Than Participants: samples
Groups:
- Cohort A (Venipuncture/SST); Cohort A (Tasso+™/SST): Samples centrifuged/aliquoted after arrival at central lab.
  Tasso+™: The Tasso+™ blood collection kit is a collection device (called the Tasso+™) and a capillary collection tube that allows for the storage of the blood in a liquid format in different matrices.
- Cohort B (Venipuncture/SST); Cohort B (Tasso+™/SST): Samples centrifuged/aliquoted at collection Site before shipment to central lab.
  Tasso+™: The Tasso+™ blood collection kit is a collection device (called the Tasso+™) and a capillary collection tube that allows for the storage of the blood in a liquid format in different matrices.
Arm/Group | Cohort A (Venipuncture/SST) | Cohort A (Tasso+™/SST) | Cohort B (Venipuncture/SST) | Cohort B (Tasso+™/SST)
Number analyzed (Participants) | 132 | 122 | 66 | 60
Number analyzed (samples) | 132 | 122 | 66 | 60
mmol/L | 139.9 (4.12) | 137.6 (8.2) | 139.7 (2.1) | 138.2 (1.82)
Statistical Analysis 1: Comparison: Cohort A (Venipuncture/SST) vs Cohort A (Tasso+™/SST); Test type: Other — Pearson's correlation coefficient were computed to quantify the strength of the direction of the linear relationship between the venipuncture collection and the Tasso+™ collection at Day 1 for each cohort for SARS-CoV-2 serology. Contingency correlation coefficient was computed to estimate the extent of the relationship between the venipuncture collection and the Tasso+™ collection at Day 1 for each cohort for each chemistry analytes; Correlation Contingency Coefficient = 0.05
Statistical Analysis 2: Comparison: Cohort B (Venipuncture/SST) vs Cohort B (Tasso+™/SST); Test type: Other — [test comment as in outcome 9, analysis 1]; Correlation Contingency Coefficient = 0.59

10. Primary Outcome: Assess the Reliability of Tasso+™
Description: Percentage of Tasso+™ device failure
Time Frame: Day 1
Population: as for outcome 1
Measure: Count of Units; unit: Devices
Units Other Than Participants: Devices
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 133 | 66 | 199
Number analyzed (Devices) | 133 | 66 | 199
Devices
  Device failure due to faulty mechanism | 2 | 2 | 4
  Device failure due to user error | 1 | 1 | 2
  No device failure | 130 | 63 | 193

11. Primary Outcome: To Assess the Reliability of Tasso+™
Description: Percentage of Tasso+™ device failure
Time Frame: Day 29
Population: as for outcome 2
Measure: Count of Units; unit: Devices
Units Other Than Participants: Devices
Arm/Group | Total
Number analyzed (Participants) | 172
Number analyzed (Devices) | 172
Devices
  Device failure due to faulty mechanism | 8
  Device failure due to user error | 0
  No Device Failures | 164

12. Primary Outcome: Assess the Reliability of Tasso+™
Description: Percentage of Tasso+™ device failure
Time Frame: Day 57
Population: as for outcome 3
Measure: Count of Units; unit: Devices
Units Other Than Participants: Devices
Arm/Group | Total
Number analyzed (Participants) | 168
Number analyzed (Devices) | 168
Devices
  Device failure due to faulty mechanism | 8
  Device failure due to user error | 2
  No device failures | 158

13. Primary Outcome: Assess the Testing Accuracy of Tasso+™ as Compared to Samples Collected Via Venipuncture for Potassium
Description: Correlation of potassium between venipuncture and Tasso+™/SST samples for each cohort
Time Frame: Day 1
Population: Full analysis
Measure: Mean (Standard Deviation); unit: mmol/L
Units Other Than Participants: samples
Arm/Group | Cohort A (Venipuncture/SST) | Cohort A (Tasso+™/SST) | Cohort B (Venipuncture/SST) | Cohort B (Tasso+™/SST)
Number analyzed (Participants) | 132 | 122 | 66 | 60
Number analyzed (samples) | 132 | 122 | 66 | 60
mmol/L | 4.31 (0.51) | 6.89 (1.8) | 4.42 (0.44) | 4.65 (1.07)
Statistical Analysis 1: Comparison: Cohort A (Venipuncture/SST) vs Cohort A (Tasso+™/SST); Test type: Other — [test comment as in outcome 9, analysis 1]; Correlation Contingency Coefficient = -0.05
Statistical Analysis 2: Comparison: Cohort B (Venipuncture/SST) vs Cohort B (Tasso+™/SST); Test type: Other — [test comment as in outcome 9, analysis 1]; Correlation Contingency Coefficient = 0.22

14. Primary Outcome: Assess the Testing Accuracy of Tasso+™ as Compared to Samples Collected Via Venipuncture for Chloride
Description: Correlation of chloride between venipuncture and Tasso+™/SST samples for each cohort
Time Frame: Day 1
Population: Full analysis
Measure: Mean (Standard Deviation); unit: mmol/L
Units Other Than Participants: samples
Arm/Group | Cohort A (Venipuncture/SST) | Cohort A (Tasso+™/SST) | Cohort B (Venipuncture/SST) | Cohort B (Tasso+™/SST)
Number analyzed (Participants) | 132 | 122 | 66 | 60
Number analyzed (samples) | 132 | 122 | 66 | 60
mmol/L | 105.8 (2.48) | 104.2 (3.7) | 106.3 (2.06) | 108.7 (2.59)
Statistical Analysis 1: Comparison: Cohort A (Venipuncture/SST) vs Cohort A (Tasso+™/SST); Test type: Other — [test comment as in outcome 9, analysis 1]; Correlation Contingency Coefficient = 0.54
Statistical Analysis 2: Comparison: Cohort B (Venipuncture/SST) vs Cohort B (Tasso+™/SST); Test type: Other — [test comment as in outcome 9, analysis 1]; Correlation Contingency Coefficient = 0.82

15. Primary Outcome: Assess the Testing Accuracy of Tasso+™ as Compared to Samples Collected Via Venipuncture for Creatinine
Description: Correlation of creatinine between venipuncture and Tasso+™/SST samples for each cohort
Time Frame: Day 1
Population: Full analysis
Measure: Mean (Standard Deviation); unit: μmol/L
Units Other Than Participants: samples
Arm/Group | Cohort A (Venipuncture/SST) | Cohort A (Tasso+™/SST) | Cohort B (Venipuncture/SST) | Cohort B (Tasso+™/SST)
Number analyzed (Participants) | 132 | 122 | 66 | 60
Number analyzed (samples) | 132 | 122 | 66 | 60
μmol/L | 71.37 (34.9) | 64.27 (36.03) | 71.67 (24.78) | 67.15 (26.1)
Statistical Analysis 1: Comparison: Cohort A (Venipuncture/SST) vs Cohort A (Tasso+™/SST); Test type: Other — [test comment as in outcome 9, analysis 1]; Correlation Contingency Coefficient = 0.96
Statistical Analysis 2: Comparison: Cohort B (Venipuncture/SST) vs Cohort B (Tasso+™/SST); Test type: Other — [test comment as in outcome 9, analysis 1]; Correlation Contingency Coefficient = 0.99

16. Primary Outcome: Assess the Testing Accuracy of Tasso+™ as Compared to Samples Collected Via Venipuncture for Glucose
Description: Correlation of glucose between venipuncture and Tasso+™/SST samples for each cohort
Time Frame: Day 1
Population: Full analysis
Measure: Mean (Standard Deviation); unit: mmol/L
Units Other Than Participants: samples
Arm/Group | Cohort A (Venipuncture/SST) | Cohort A (Tasso+™/SST) | Cohort B (Venipuncture/SST) | Cohort B (Tasso+™/SST)
Number analyzed (Participants) | 132 | 121 | 66 | 59
Number analyzed (samples) | 132 | 121 | 66 | 59
mmol/L | 5.33 (1.63) | 1.38 (1.72) | 5.23 (1.92) | 5.58 (2.17)
Statistical Analysis 1: Comparison: Cohort A (Venipuncture/SST) vs Cohort A (Tasso+™/SST); Test type: Other — [test comment as in outcome 9, analysis 1]; Correlation Contingency Coefficient = 0.63
Statistical Analysis 2: Comparison: Cohort B (Venipuncture/SST) vs Cohort B (Tasso+™/SST); Test type: Other — [test comment as in outcome 9, analysis 1]; Correlation Contingency Coefficient = 0.95

17. Primary Outcome: Assess the Testing Accuracy of Tasso+™ as Compared to Samples Collected Via Venipuncture for Phosphate
Description: Correlation of phosphate between venipuncture and Tasso+™/SST samples for each cohort
Time Frame: Day 1
Population: Full analysis
Measure: Mean (Standard Deviation); unit: mmol/L
Units Other Than Participants: samples
Arm/Group | Cohort A (Venipuncture/SST) | Cohort A (Tasso+™/SST) | Cohort B (Venipuncture/SST) | Cohort B (Tasso+™/SST)
Number analyzed (Participants) | 132 | 122 | 66 | 60
Number analyzed (samples) | 132 | 122 | 66 | 60
mmol/L | 1.1 (0.18) | 1.98 (1.87) | 1.1 (0.17) | 1.08 (0.16)
Statistical Analysis 1: Comparison: Cohort A (Venipuncture/SST) vs Cohort A (Tasso+™/SST); Test type: Other — [test comment as in outcome 9, analysis 1]; Correlation Contingency Coefficient = 0.03
Statistical Analysis 2: Comparison: Cohort B (Venipuncture/SST) vs Cohort B (Tasso+™/SST); Test type: Other — [test comment as in outcome 9, analysis 1]; Correlation Contingency Coefficient = 0.95

18. Primary Outcome: Assess the Testing Accuracy of Tasso+™ as Compared to Samples Collected Via Venipuncture for Urate
Description: Correlation of urate between venipuncture and Tasso+™/SST samples for each cohort
Time Frame: Day 1
Population: Full analysis
Measure: Mean (Standard Deviation); unit: mmol/L
Units Other Than Participants: samples
Arm/Group | Cohort A (Venipuncture/SST) | Cohort A (Tasso+™/SST) | Cohort B (Venipuncture/SST) | Cohort B (Tasso+™/SST)
Number analyzed (Participants) | 132 | 120 | 66 | 59
Number analyzed (samples) | 132 | 120 | 66 | 59
mmol/L | 0.3 (0.08) | 0.28 (0.09) | 0.3 (0.1) | 0.29 (0.09)
Statistical Analysis 1: Comparison: Cohort A (Venipuncture/SST) vs Cohort A (Tasso+™/SST); Test type: Other — [test comment as in outcome 9, analysis 1]; Correlation Contingency Coefficient = 0.85
Statistical Analysis 2: Comparison: Cohort B (Venipuncture/SST) vs Cohort B (Tasso+™/SST); Test type: Other — [test comment as in outcome 9, analysis 1]; Correlation Contingency Coefficient = 0.97

19. Primary Outcome: Assess the Testing Accuracy of Tasso+™ as Compared to Samples Collected Via Venipuncture for C-reactive Protein
Description: Correlation of C-reactive protein between venipuncture and Tasso+™/SST samples for each cohort
Time Frame: Day 1
Population: Full analysis
Measure: Mean (Standard Deviation); unit: mg/L
Units Other Than Participants: samples
Arm/Group | Cohort A (Venipuncture/SST) | Cohort A (Tasso+™/SST) | Cohort B (Venipuncture/SST) | Cohort B (Tasso+™/SST)
Number analyzed (Participants) | 132 | 121 | 66 | 60
Number analyzed (samples) | 132 | 121 | 66 | 60
mg/L | 5.19 (12.47) | 4.98 (11.54) | 4.34 (7.89) | 4.44 (8.06)
Statistical Analysis 1: Comparison: Cohort A (Venipuncture/SST) vs Cohort A (Tasso+™/SST); Test type: Other — [test comment as in outcome 9, analysis 1]; Correlation Contingency Coefficient = 0.99
Statistical Analysis 2: Comparison: Cohort B (Venipuncture/SST) vs Cohort B (Tasso+™/SST); Test type: Other — [test comment as in outcome 9, analysis 1]; Correlation Contingency Coefficient = 1.0

20. Secondary Outcome: To Evaluate Tasso+™ User Experience (Safety)
Description: Percentage of eligible participants who experience solicited local adverse events (AEs) including pain, tenderness, redness, swelling, or bruising within 7 days of Tasso+™ administration
Time Frame: Within 7 days of Tasso+™ administration
Population: Full analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 134 | 66 | 200
Participants | 71 | 39 | 110

21. Secondary Outcome: To Evaluate Tasso+™ User Experience (Safety)
Description: Percentage of eligible subjects who experienced unsolicited AEs within 28 days of Tasso+™ administration
Time Frame: Day 29
Population: Full analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 134 | 66 | 200
Participants | 15 | 13 | 28

22. Secondary Outcome: To Evaluate Tasso+™ User Experience (Safety)
Description: Percentage of eligible subjects who experienced a related Grade 3 AE, a related Grade 4 AE, a related AE leading to study discontinuation, or a related SAE within 28 days of Tasso+™ administration
Time Frame: Day 29
Population: Full analysis
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 134 | 66 | 200
percentage of participants
  Subjects experienced a related Grade 3 AE | 0 | 0 | 0
  Subjects experienced a related Grade 4 AE | 0 | 0 | 0
  Subjects experienced a related AE leading to discontinuation | 0 | 0 | 0
  Subjects experienced a related SAE | 0 | 0 | 0

23. Secondary Outcome: To Evaluate Tasso+™ User Experience (Tolerability)
Description: Percentage of eligible participants who complete last Tasso+™ administration (Day 57)
Time Frame: Day 57
Population: Full analysis including all subjects (Cohorts A and B) administered Tasso+™ on Day 57. The analysis population in the Day 57 endpoints includes all subjects regardless of cohort. Completion of Tasso+™ administration is not cohort specific as it was pre-specified to collect and report as a total for both cohorts.
Measure: Count of Participants; unit: Participants
Arm/Group | Total
Number analyzed (Participants) | 200
Participants | 153

24. Secondary Outcome: To Evaluate Tasso+™ User Experience (Usability)
Description: Ease of use as assessed by the participant completing the Tasso questionnaire immediately following administration
Time Frame: Day 1
Population: Full analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 134 | 66 | 200
Participants
  Questionnaire how easy was the Tasso+™ device to use? Score: 1 (Easy) | 100 | 38 | 138
  Questionnaire how easy was the Tasso+™ device to use? Score: 2 | 13 | 12 | 25
  Questionnaire how easy was the Tasso+™ device to use? Score: 3 | 0 | 3 | 6
  Questionnaire how easy was the Tasso+™ device to use? Score: 4 | 4 | 1 | 3
  Questionnaire how easy was the Tasso+™ device to use? Score: 5 (Difficult) | 3 | 3 | 6
  Questionnaire results unknown | 14 | 9 | 22

25. Secondary Outcome: To Evaluate Tasso+™ User Experience (Usability)
Description: Ease of use as assessed by the participant completing the Tasso questionnaire immediately following administration
Time Frame: Day 29
Population: Full analysis including all subjects (Cohorts A and B) administered Tasso+™ on Day 29. The analysis population in the Day 29 endpoints includes all subjects regardless of cohort. Ease of use as assessed by the participant completing the Tasso questionnaire immediately following administration is not cohort specific as it was pre-specified to collect and report as a total for both cohorts. .
Measure: Count of Participants; unit: Participants
Arm/Group | Total
Number analyzed (Participants) | 200
Participants
  Questionnaire how easy was the Tasso+™ device to use? Score: 1 (Easy) | 130
  Questionnaire how easy was the Tasso+™ device to use? Score: 2 | 11
  Questionnaire how easy was the Tasso+™ device to use? Score: 3 | 5
  Questionnaire how easy was the Tasso+™ device to use? Score: 4 | 2
  Questionnaire how easy was the Tasso+™ device to use? Score: 5 (Difficult) | 6
  Questionnaire results unknown | 46

26. Secondary Outcome: To Evaluate Tasso+™ User Experience (Usability)
Description: Ease of use as assessed by the participant completing the Tasso questionnaire immediately following administration
Time Frame: Day 57
Population: Full analysis including all subjects (Cohorts A and B) administered Tasso+™ on Day 57. The analysis population in the Day 57 endpoints includes all subjects regardless of cohort. Ease of use as assessed by the participant completing the Tasso questionnaire immediately following administration is not cohort specific as it was pre-specified to collect and report as a total for both cohorts.
Measure: Count of Participants; unit: Participants
Arm/Group | Total
Number analyzed (Participants) | 200
Participants
  Questionnaire how easy was the Tasso+™ device to use? Score: 1 (Easy) | 137
  Questionnaire how easy was the Tasso+™ device to use? Score: 2 | 8
  Questionnaire how easy was the Tasso+™ device to use? Score: 3 | 2
  Questionnaire how easy was the Tasso+™ device to use? Score: 4 | 3
  Questionnaire how easy was the Tasso+™ device to use? Score: 5 (Difficult) | 5
  Questionnaire results unknown | 45

27. Secondary Outcome: To Evaluate Tasso+™ User Experience (Usability)
Description: Willingness to use the Tasso device was assessed by the participant completing the Tasso questionnaire
Time Frame: Day 85
Population: Full analysis including all subjects (cohorts A and B) as the willingness to use the Tasso device is not cohort specific as it was pre-specified to collect and report as a total for both cohorts.
Measure: Count of Participants; unit: Participants
Arm/Group | Total
Number analyzed (Participants) | 200
Participants
  How often would you be willing to provide a blood sample using the Tasso+™ device? 1 per year | 13
  How often would you be willing to provide a blood sample using the Tasso+™ device? 1 per month | 32
  How often would you be willing to provide a blood sample using the Tasso+™ device? 1 per week | 17
  How often would you be willing to provide a blood sample using the Tasso+™ device? 1 per day | 7
  How often would you be willing to provide a blood sample using the Tasso+™ device? Never | 3
  How often would you be willing to provide a blood sample using the Tasso+™ device? As needed | 97
  Questionnaire results unknown | 31

28. Secondary Outcome: To Perform Surveillance for SARS-CoV-2 Infection
Description: Percentage of eligible participants with a positive nasopharyngeal swab for SARS-CoV-2 polymerase chain reaction (PCR) on Day 1
Time Frame: Day 1
Population: Full analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 134 | 66 | 200
Participants | 3 | 1 | 4

29. Secondary Outcome: To Perform Surveillance for SARS-CoV-2 Infection
Description: Percentage of eligible participants seroconverting to SARS-CoV-2 between Days 1 and 57
Time Frame: Between Days 1 and 57
Population: Full analysis including all subjects (cohorts A and B) as Percentage of eligible participants seroconverting to SARS-CoV-2 between Days 1 and 57 is not cohort specific as it was pre-specified to collect and report as a total for both cohorts.
Measure: Count of Participants; unit: Participants
Arm/Group | Total
Number analyzed (Participants) | 200
Participants | 0

30. Secondary Outcome: To Evaluate Tasso+™ User Experience (Usability)
Description: Willingness to use the Tasso device was assessed by the participant completing the Tasso questionnaire
Time Frame: Day 29
Population: Full analysis including all subjects (Cohorts A and B) administered Tasso+™ on Day 29. The analysis population in the Day 29 endpoints includes all subjects regardless of cohort as this outcome is not cohort specific as it was pre-specified to collect and report as a total for both cohorts.
Measure: Count of Participants; unit: Participants
Arm/Group | Total
Number analyzed (Participants) | 200
Participants
  How often would you be willing to provide a blood sample using the Tasso+™ device? 1 per year | 6
  How often would you be willing to provide a blood sample using the Tasso+™ device? 1 per month | 24
  How often would you be willing to provide a blood sample using the Tasso+™ device? 1 per week | 24
  How often would you be willing to provide a blood sample using the Tasso+™ device? 1 per day | 8
  How often would you be willing to provide a blood sample using the Tasso+™ device? Never | 1
  How often would you be willing to provide a blood sample using the Tasso+™ device? As needed | 91
  Questionnaire results unknown | 46

31. Secondary Outcome: To Evaluate Tasso+™ User Experience (Usability)
Description: Willingness to use the Tasso device was assessed by the participant completing the Tasso questionnaire
Time Frame: Day 57
Population: Full analysis including all subjects (Cohorts A and B) administered Tasso+™ on Day 57. The analysis population in the Day 57 endpoints includes all subjects regardless of cohort. Willingness to use the Tasso device is not cohort specific as it was pre-specified to collect and report as a total for both cohorts.
Measure: Count of Participants; unit: Participants
Arm/Group | Total
Number analyzed (Participants) | 200
Participants
  How often would you be willing to provide a blood sample using the Tasso+™ device? 1 per year | 9
  How often would you be willing to provide a blood sample using the Tasso+™ device? 1 per month | 22
  How often would you be willing to provide a blood sample using the Tasso+™ device? 1 per week | 22
  How often would you be willing to provide a blood sample using the Tasso+™ device? 1 per day | 7
  How often would you be willing to provide a blood sample using the Tasso+™ device? Never | 0
  How often would you be willing to provide a blood sample using the Tasso+™ device? As needed | 95
  Questionnaire results unknown | 45

32. Secondary Outcome: To Evaluate Tasso+™ User Experience (Usability)
Description: Willingness to use the Tasso device was assessed by the participant completing the Tasso questionnaire
Time Frame: Day 1
Population: Full analysis including all subjects (Cohorts A and B) administered Tasso+™ on Day 1. The analysis population in the Day 1endpoints includes all subjects regardless of cohort as it was pre-specified to collect and report as a total for both cohorts.
Measure: Count of Participants; unit: Participants
Arm/Group | Total
Number analyzed (Participants) | 200
Participants
  How often would you be willing to provide a blood sample using the Tasso+™ device? 1 per year | 8
  How often would you be willing to provide a blood sample using the Tasso+™ device? 1 per month | 25
  How often would you be willing to provide a blood sample using the Tasso+™ device? 1 per week | 22
  How often would you be willing to provide a blood sample using the Tasso+™ device? 1 per day | 16
  How often would you be willing to provide a blood sample using the Tasso+™ device? Never | 2
  How often would you be willing to provide a blood sample using the Tasso+™ device? As needed | 104
  Questionnaire results unknown | 23

33. Secondary Outcome: To Evaluate Tasso+™ User Experience (Usability)
Description: Preferred method for future blood sampling was assessed by the participant completing the Tasso questionnaire
Time Frame: Day 85
Population: Full analysis including all subjects (Cohorts A and B) administered Tasso+™ on Day 85. The analysis population in the Day 85 endpoints includes all subjects regardless of cohort. Determining the method for future blood sampling by the participant is not cohort specific as both cohorts had blood collected using the Tasso device and the venipuncture method and it was pre-specified to collect and report as a total for both cohorts.
Measure: Count of Participants; unit: Participants
Arm/Group | Total
Number analyzed (Participants) | 200
Participants
  How would you prefer future blood sampling? Tasso+™ device self-applied at home | 134
  How would you prefer future blood sampling? Tasso+™ device applied at doctor's office or a lab | 16
  How would you prefer future blood sampling? Venipuncture at doctor's office or a lab | 10
  How would you prefer future blood sampling? Finger stick device self-applied at home | 5
  How would you prefer future blood sampling? Finger stick device applied at doctor's office or a lab | 4
  Questionnaire results unknown | 31

34. Other Pre Specified Outcome: To Evaluate the Impact of Prior Training on Subsequent Tasso+™ Administrations and Sample Integrity
Description: Percentage of Tasso+™/SST samples collected that are with adequate volume and without moderate or gross hemolysis between patients who requested proctor-supported and those who did not request proctor-supported for the usage of Tasso+™ on Day 57
Time Frame: Day 57
Population: Per the SAP, the Per-Protocol Set will include all participants who successfully completed at least five Tasso+™ administrations and do not have any important protocol deviations. This analysis set will be used for sensitivity analyses.
Measure: Number; unit: percentage of samples
Units Other Than Participants: samples
Groups:
- Proctor Supported Tasso+™ Administrations: Subjects from either cohort who requested proctor supported Tasso+™ Administration on Day 57
- Proctor Unsupported Tasso+™ Administrations: Subjects from either cohort who did not requested proctor supported Tasso+™ Administration on Day 57
- Total: Subjects from either cohort who did and did not requested proctor supported Tasso+™ Administration on Day 57
Arm/Group | Proctor Supported Tasso+™ Administrations | Proctor Unsupported Tasso+™ Administrations | Total
Number analyzed (Participants) | 16 | 69 | 85
Number analyzed (samples) | 16 | 69 | 85
percentage of samples | 41.2 | 48.6 | 47.2

35. Other Pre Specified Outcome: To Evaluate the Impact of Prior Training on Subsequent Tasso+™ Administrations and Sample Integrity
Description: Percentage of Tasso+™/EDTA samples collected that are with adequate volume and without moderate or gross hemolysis between patients who requested proctor-supported and those who did not request proctor-supported for the usage of Tasso+™ on Day 57
Time Frame: Day 57
Population: as for outcome 34
Measure: Number; unit: percentage of samples
Units Other Than Participants: samples
Arm/Group | Proctor Supported Tasso+™ Administrations | Proctor Unsupported Tasso+™ Administrations | Total
Number analyzed (Participants) | 16 | 67 | 83
Number analyzed (samples) | 16 | 67 | 83
percentage of samples | 0 | 6.9 | 5.6

36. Other Pre Specified Outcome: To Evaluate the Impact of Prior Training on Subsequent Tasso+™ Administrations and Reliability
Description: Percentage of Tasso+™ device failure between patients who requested proctor-supported and those who did not request proctor-supported for the usage of Tasso+™ on Day 57
Time Frame: Day 57
Population: Per-Protocol
Measure: Number; unit: percentage of device failures
Units Other Than Participants: devices
Arm/Group | Proctor Supported Tasso+™ Administrations | Proctor Unsupported Tasso+™ Administrations | Total
Number analyzed (Participants) | 17 | 72 | 89
Number analyzed (devices) | 17 | 72 | 89
percentage of device failures
  Device failure due to faulty mechanism | 11.8 | 2.8 | 4.5
  Device failure due to user error | 0 | 0 | 0

37. Other Pre Specified Outcome: To Evaluate the Impact of Prior Training on Subsequent Tasso+™ Administrations and Safety
Description: Percentage of subjects with solicited local AEs within 7 days of Tasso+™ administration on Day 57 between patients who requested proctor-supported and those who did not request proctor-supported for the usage of Tasso+™
Time Frame: Within 7 days of Tasso+™ administration on Day 57, up to a maximum of 64 days
Population: Per-Protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Proctor Supported Tasso+™ Administrations | Proctor Unsupported Tasso+™ Administrations | Total
Number analyzed (Participants) | 17 | 72 | 89
Participants
  Solicited local AEs | 7 | 30 | 37
  No solicited local AEs | 10 | 42 | 52

38. Other Pre Specified Outcome: To Evaluate the Impact of Prior Training on Subsequent Tasso+™ Administrations and Safety
Description: Percentage of subjects with unsolicited AEs, related Grade 3 AE, related Grade 4 AE, related AE leading to discontinuation, or related SAE within 28 days of Tasso+™ administration on between patients who requested proctor-supported and those who did not request proctor-supported for the usage of Tasso+™ on Day 57
Time Frame: Within 28 days of Tasso+™ administration on Day 57, up to Day 85
Population: Per-Protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Proctor Supported Tasso+™ Administrations | Proctor Unsupported Tasso+™ Administrations | Total
Number analyzed (Participants) | 17 | 72 | 89
Participants
  Subjects experienced unsolicited AEs | 1 | 0 | 1
  Subjects experienced a related Grade 3 AE | 0 | 0 | 0
  Subjects experienced a related Grade 4 AE | 0 | 0 | 0
  Subjects experienced a related AE leading to discontinuation | 0 | 0 | 0
  Subjects experienced a related SAE | 0 | 0 | 0
  No unsolicited AEs, related Grade 3 AE, Grade 4 AE, AE leading to discontinuation, or SAE | 16 | 72 | 88

39. Other Pre Specified Outcome: To Evaluate the Impact of Prior Training on Subsequent Tasso+™ Administrations and Usability
Description: Ease of use as assessed by the participant completing the Tasso questionnaire immediately following administration
Time Frame: Day 57
Population: Per-Protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Proctor Supported Tasso+™ Administrations | Proctor Unsupported Tasso+™ Administrations | Total
Number analyzed (Participants) | 17 | 72 | 89
Participants
  Questionnaire how easy was the Tasso+™ device to use? Score: 1 (Easy) | 13 | 65 | 78
  Questionnaire how easy was the Tasso+™ device to use? Score: 2 | 2 | 4 | 6
  Questionnaire how easy was the Tasso+™ device to use? Score: 3 | 0 | 0 | 0
  Questionnaire how easy was the Tasso+™ device to use? Score: 4 | 2 | 0 | 3
  Questionnaire how easy was the Tasso+™ device to use? Score: 5 (Difficult) | 0 | 3 | 2
  Questionnaire results unknown | 0 | 0 | 0

40. Other Pre Specified Outcome: To Evaluate the Impact of Prior Training on Subsequent Tasso+™ Administrations and Usability
Description: Willingness to use the Tasso device was assessed by the participant completing the Tasso questionnaire
Time Frame: Day 57
Population: Per-Protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Proctor Supported Tasso+™ Administrations | Proctor Unsupported Tasso+™ Administrations | Total
Number analyzed (Participants) | 17 | 72 | 89
Participants
  How often would you be willing to provide a blood sample using the Tasso+™ device? 1 per year | 1 | 3 | 4
  How often would you be willing to provide a blood sample using the Tasso+™ device? 1 per month | 0 | 13 | 13
  How often would you be willing to provide a blood sample using the Tasso+™ device? 1 per week | 3 | 9 | 12
  How often would you be willing to provide a blood sample using the Tasso+™ device? 1 per day | 0 | 3 | 3
  How often would you be willing to provide a blood sample using the Tasso+™ device? None | 0 | 0 | 0
  How often would you be willing to provide a blood sample using the Tasso+™ device? As needed | 0 | 0 | 0
  Questionnaire results unknown | 13 | 44 | 57

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Cohort A | Cohort B | Total
All-Cause Mortality (participants affected / at risk) | 0/134 | 0/66 | 0/200
Serious Adverse Events (participants affected / at risk) | 0/134 | 0/66 | 0/200
Other Adverse Events (participants affected / at risk) | 76/134 | 40/66 | 116/200
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=134) | Cohort B (N=66) | Total (N=200)
Administration site pain (General disorders) | 43 | 30 | 73
Administration site scar (General disorders) | 46 | 24 | 70
Administration site erythema (General disorders) | 32 | 19 | 51
Administration site swelling (General disorders) | 21 | 12 | 33
Administration site bruise (General disorders) | 16 | 10 | 26
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 6
Headache (Nervous system disorders) | 1 | 3 | 4
Chills (General disorders) | 1 | 2 | 3
Administration site pruritus (General disorders) | 2 | 1 | 3
Fatigue (General disorders) | 1 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 2 | 3
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2
Acute sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 1
Ear infection (Infections and infestations) | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 1
Norovirus infection (Infections and infestations) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2025-01-17): https://cdn.clinicaltrials.gov/large-docs/66/NCT06507566/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT06507566/SAP_001.pdf